CLINICAL TRIAL: NCT01229904
Title: Guitars for Vets: Evaluating Psychological Outcome of a Novel Music Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPO 10-075
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2011-07

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): patients with PTSD are randomized to either entering immediately a 6 week treatment with music therapy, or being in the delay group that enters the treatment arm after 6 weeks. This is a delayed entry RCT.
  Interventions: Behavioral: music therapy with guitar lessons

INTERVENTIONS:
Behavioral: music therapy with guitar lessons — The treatment is a 6 week music therapy intervention. Subjects receive 1 hour individual lesson and a 1 hour group session weekly for 6 weeks. they are given a guitar following completion of the study

SUMMARY:
Post traumatic Stress disorder (PTSD) is a common condition for persons who have served in the Armed services during combat or deployment. Treatments include medications, cognitive behavioral therapy, and other social support mechanisms.

Our aim in this project is to critically evaluate the effects of a novel music therapy intervention on the symptoms of PTSD. Estimates developed by the Global Burden of Disease Study reveal that mental illness accounts for over 15% of the burden of disease on health and productivity in established market economies--more than the disease burden caused by all cancers combined.[1] Perhaps no industry has had the burden of mental disorders affect its labor force as severely and pervasively as the Armed Forces.

Post-Traumatic Stress Disorder (PTSD) is a common sequelae of severe emotional trauma that is often associated with combat exposure. The condition has been well documented in returning soldiers and is characterized by recurrent and distressing thoughts and feelings related to the trauma, persistent avoidance of reminders of the trauma, and increased arousal that disturbs sleep, concentration, and the ability to modulate anger. Persons suffering from PTSD often have difficulty relating to others, leading to loneliness and isolation, which further intensifies their psychiatric symptoms. Current treatment options for PTSD include psychotherapy, medication management, or a combination of those. Although these treatments have been shown to be effective, returning soldiers are often hesitant to seek and adhere to mental health therapies. PTSD-related avoidance, including difficulty trusting, may serve as a barrier to seeking or completing treatments. Furthermore, some PTSD medications have unacceptable side-effects in some individuals. The need is great, therefore, to identify and promote safe, effective strategies for self-management of PTSD among Veterans.

DETAILED DESCRIPTION:
Background:

Post traumatic Stress disorder (PTSD) is a common condition for persons who have served in the Armed services during combat or deployment. Treatments include medications, cognitive behavioral therapy, and other social support mechanisms.

Our aim in this project is to critically evaluate the effects of a novel music therapy intervention on the symptoms of PTSD. Estimates developed by the Global Burden of Disease Study reveal that mental illness accounts for over 15% of the burden of disease on health and productivity in established market economies--more than the disease burden caused by all cancers combined.[1] Perhaps no industry has had the burden of mental disorders affect its labor force as severely and pervasively as the Armed Forces.

Post-Traumatic Stress Disorder (PTSD) is a common sequelae of severe emotional trauma that is often associated with combat exposure. The condition has been well documented in returning soldiers and is characterized by recurrent and distressing thoughts and feelings related to the trauma, persistent avoidance of reminders of the trauma, and increased arousal that disturbs sleep, concentration, and the ability to modulate anger. Persons suffering from PTSD often have difficulty relating to others, leading to loneliness and isolation, which further intensifies their psychiatric symptoms. Current treatment options for PTSD include psychotherapy, medication management, or a combination of those. Although these treatments have been shown to be effective, returning soldiers are often hesitant to seek and adhere to mental health therapies. PTSD-related avoidance, including difficulty trusting, may serve as a barrier to seeking or completing treatments. Furthermore, some PTSD medications have unacceptable side-effects in some individuals. The need is great, therefore, to identify and promote safe, effective strategies for self-management of PTSD among Veterans.

Objectives:

The objective was to assess the effectiveness of a novel music therapy on ammelorating the effects of PTSD. Specifically a 6 week guitar training program under the direction of seasoned instructors through a partnership with Guitars for Vets was assessed before and after intervention.

Methods:

In this trial we recruited veterans in the Milwaukee region and the Zablocki VA Medical Center with significant PTSD symptoms. Forty subjects were recruited and randomized to either an immediate entry or a 6 week delayed entry group. Both groups received the intervention, but the delayed group received it after a 6 week period.

Each subject received a guitar that they keep after the study, music, supplies and instructions. They each had an hour of individual training each week and a weekly group instruction session.

Status:

The data collection and analyses are complete, we are writing the final manuscript. In addition, we submitted a grant for a multicenter MERIT funded project this past June. Unfortunately it will not be funded. We plan to resubmit at the next cycle.

ELIGIBILITY:
Inclusion Criteria:

Veterans in the Zablocki VA catchment area with symptomatic post traumatic stress disorder

Exclusion Criteria:

Current involvement in intense treatment for a psychiatric illness or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress disorder Checklist (PCL) | after 6 weeks of intervention with music training

SECONDARY OUTCOMES:
depression, social participation, wellness | after 6 weeks of intervention with music training

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R. Dillingham, MD MS, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States